CLINICAL TRIAL: NCT05387967
Title: Safety and Tolerability of Sacubitril/Valsartan in Heart Failure Patient With Reduced Ejection Fraction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Cardiovascular Diseases, Pakistan (Other)
Responsible Party: Principal Investigator, Dr. Muhammad Nauman Khan, Assistant Professor of Cardiology, National Institute of Cardiovascular Diseases, Pakistan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ERC-05/2020
Record Dates: First submitted 2022-05-13; First posted 2022-05-24 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Heart Failure, Systolic
MeSH Terms: conditions — Heart Failure, Systolic | interventions — sacubitril and valsartan sodium hydrate drug combination; Angiotensin Receptor Antagonists

STUDY DESIGN:
Intervention Model Description: Open label non-randomized clinical trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): All the recruited patients were prescribed Sacubitril/Valsartan at a starting dose of 50 (24/26) mg BID which was up-titrated, over the period of initial 6 weeks, to the maximum tolerated dose up to 200 (97/103) mg BID and further followed for a total of 12 weeks.
  Interventions: Drug: Sacubitril/valsartan

INTERVENTIONS:
Drug: Sacubitril/valsartan — All the recruited patients were prescribed Sacubitril/Valsartan at a starting dose of 50 (24/26) mg BID which was up-titrated, over the period of initial 6 weeks, to the maximum tolerated dose up to 200 (97/103) mg BID and further followed for a total of 12 weeks.
  Other Names: Angiotensin receptor blocker and neprilysin inhibitor (ARNI)

SUMMARY:
This proof-of-concept, open-label non-randomized clinical trial was conducted at a tertiary care cardiac center in Karachi, Pakistan. Patients with HFrEF were prescribed Sacubitril/Valsartan and followed for 12 weeks for the assessment of safety and tolerability. Safety measures included incidence of hypotension, renal dysfunction, hyperkalemia, and angioedema

DETAILED DESCRIPTION:
A required number of consecutive patients meeting the inclusion criteria were recruited for this study. After written informed consent patient demographic and baseline clinical characteristics were obtained. Inclusion criteria for the study were either gender between 18 to 80 years of age, diagnosed with congestive heart failure (CHF) with NYHA class II-IV, and LVEF ≤ 40%. Pre-inclusion safety parameters were patients who were stable on any dose of beta-blockers, angiotensin-converting enzyme inhibitor (ACEI) or angiotensin receptor blocker (ARB) prior to enrolment in the study. Patients with a baseline diagnosis of Hyperkalemia, hypotension, renal dysfunction, and a history of hypersensitivity to the active substances, Sacubitril/Valsartan, or to any of the excipients or drugs of similar chemical classes were excluded from the study.

All the recruited patients were prescribed Sacubitril/Valsartan 100mg/200mg twice a day (BID) for 6 weeks. A weekly telephonic follow-up was made to assess the patient's medication adherence level using the Dose-Nonadherence scale. All the patients were kept under a close follow-up for 6 weeks period and at the end of 12 weeks of medication, the safety and tolerability outcomes were assessed as per the operational definition.

ELIGIBILITY:
Inclusion Criteria:

* Either gender
* between 18 to 80 years of age
* Diagnosed with Heart failure with reduced ejection fraction (HFrEF)
* New York Heart Association (NYHA) class II-IV
* Left ventricular ejection fraction (LVEF) ≤ 40%
* Stable on any dose of beta-blockers, ACEI or ARB

Exclusion Criteria:

* Refused to participate in the study
* Patients with hyperkalemia
* Patients with hypotension
* Patients with renal dysfunction
* History of hypersensitivity to the active substances, Sacubitril/Valsartan, or to any of the excipients or drugs of similar chemical classes

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Incidence of hypotension | 12 weeks
  Systolic blood pressure <90 mmHg
Incidence of renal dysfunction | 12 weeks
  estimated glomerular filtration rate (eGFR) <30 ml/min
Incidence of renal hyperkalemia | 12 weeks
  Potassium >5.2 mmol/L
Incidence of renal angioedema | 12 weeks
  Rapid edema, or swelling, of the area beneath the skin or mucosa
Frequency of tolerability | During 12 weeks
  Defined as the dose tolerated by the patients which did not require down titration or discontinuation of prescribed dose during follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Nauman Khan, FCPS, Principal Investigator — National Institute of Cardiovascular Diseases (NICVD), Karachi, Pakistan
Locations (1):
- National Institute of Cardiovascular Diseases, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Khan MN, Soomro NA, Naseeb K, Bhatti UH, Rauf R, Balouch IJ, Moazzam A, Bashir S, Ashraf T, Karim M. Safety and tolerability of Sacubitril/Valsartan in heart failure patient with reduced ejection fraction. BMC Cardiovasc Disord. 2023 Mar 13;23(1):133. doi: 10.1186/s12872-023-03070-9. PMID 36915075